CLINICAL TRIAL: NCT01234636
Title: Effects of cis9,trans11 Conjugated Linoleic Acid on Platelet Function, Markers of Haemostasis and Inflammation on Humans
Brief Title: Conjugated Linoleic Acid Supplementation Study
Acronym: CLASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RINH_1000
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Cardiovascular Disease
Keywords: Platelets; Platelet aggregation; Platelet activation; Platelet function; Light transmission aggregometry; Flow cytometry; Platelet function analyzer-100 (PFA-100); Linoleic acid, conjugated; cis9, trans11 conjugated linoleic acid; dietary supplement; short-term intervention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cis9,trans 11 CLA oil (Active Comparator): 50 volunteers on cross over design , receiving 4g/day of cis9,trans11 CLA
  Interventions: Dietary Supplement: Placebo oil
- Placebo oil (Placebo Comparator): 50 volunteers cross over design, placebo oil 4g/day
  Interventions: Dietary Supplement: Placebo oil

INTERVENTIONS:
Dietary Supplement: Placebo oil — Placebo oil of 4g/day

SUMMARY:
Cardiovascular disease is a major cause of mortality worldwide resulting in one out of three global deaths. One of the main characteristics of cardiovascular disease is impaired blood flow and increased formation of clots. Platelets are clot-forming cells responsible for prevention of bleeding. However, in disease state they may be overly activated and tend to stick to each other, promoting blood clots and blockage of vessels.

Conjugated linoleic acids (CLA) are unique fatty acids present in dairy food products and beef which would help to prevent platelets from clotting and thus help to prevent cardiovascular disease. However, the mechanisms by which those fatty acids affect platelet function are not yet fully understood. We designed a human intervention study assessing the mechanisms by which CLA beneficially affect platelet function and markers of haemostasis and inflammation in humans.

DETAILED DESCRIPTION:
Despite being trans fatty acids, dietary conjugated linoleic acids( CLA) have been associated with decreased atherogenesis, beneficial effects on insulin sensitivity , glucose and lipid profile and body composition in animal studies.Todate only few studies have studied the effects of the two individual CLA isomers on body composition , lipoprotein metabolism immune function , inflammation , insulin sensitivity and oxidative stress in humans.

A previous study revealed that both cis9,trans11 and trans10,cis12 CLA, as well as CLA mix, significantly decreased agonist-induced platelet aggregation and TxB2 production ex vivo compared with linoleic acid. No effect on agonist-induced platelet aggregation or other blood clotting parameters in healthy female volunteers was observed upon supplementation with 3.9 g/d CLA, compared with sunflower oil, but this may have been due to the low number of subjects participating in this study.

Indeed, supplementation with 13.0 g/day of CLA mix - 50:50 blend, compared with placebo oil, significantly decreased fibrinogen levels in type 2 diabetes patients, and fibrinogen and plasminogen activator inhibitor-1 levels were significantly lower upon intervention with CLA milk (4.7 g/d cis9,trans11 CLA and 0.4 g/d trans10,cis12 CLA), compared with CLA mix (2.3 g/d cis9,trans11 CLA and 2.2 g/d trans10,cis12 CLA), and lower compared with olive oil, in postmenopausal women.Thus overall evidence indicates that especially the cis9,trans11 CLA isomer may prevent platelet activation and aggregation, and possibly display anticoagulant properties. However, so far this has not been assessed in detail.

In this study we assess effects of supplementation of cis9,trans11 CLA-rich oil on platelet function by measuring not only platelet aggregation but also in vitro coagulation and platelet activation in healthy overweight humans. In addition, we examine the effects of CLA supplementation on plasma and cellular marker of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:• Healthy men and women aged 35-74 years

* blood pressure below 160/90 mmHg;
* fasting plasma glucose < 7 mmol/L;
* total cholesterol < 8 mmol/L,with cholesterol/HDL ratio < 6 and/or ASSIGN score < 20%)
* platelet count > 170x109/L
* haematocrit above 40 % for males and above 35 % for females
* haemoglobin above 130 g/L for males and above 115 g/L for females
* having a 10-20% risk for developing cardiovascular disease within the next 10 years based on the ASSIGN calculation (http://cvrisk.mvm.ed.ac.uk/index.htm) including the following factors: age, gender, number of cigarettes smoked per day, Scottish Index of Multiple Deprivation (SIMD)/postcode, systolic blood pressure, levels of total and HDL cholesterol and family history of cardiovascular disease or having at least one additional risk factor such as being over 50 years old, BMI above 25 kg/m2, elevated triglyceride levels (> 1.7 mmol/L) or elevated glucose levels (> 5.6 mmol/L);

Exclusion Criteria:Exclusion criteria Subjects are excluded if

* They are regularly taking aspirin or aspirin-containing drugs, or other anti-inflammatory drugs;
* They are taking drugs or herbal medicines known to alter platelet function or the haemostatic system in general;
* They are diagnosed with diabetes, hypertension, renal, hepatic, haematological disease or coronary heart disease;
* They are undertaking more than 6 hours vigorous exercise per week
* They are pregnant (or planning to become pregnant) or lactating;
* They have given a pint of blood for transfusion purposes within the last month;
* They have unsuitable veins for blood sampling;
* They are inability to understand the participant information sheet or inability to speak, read and understand the English language.

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change of expression of P-selectin and fibrinogen receptor activation on platelets by flow cytometry | At 2 weeks
  Using fluorescently-conjugated monoclonal antibodies and whole blood flow cytometry after ex vivo stimulation with adenosine diphosphate (ADP), thrombin receptor-activating peptide (TRAP) P-selectin expression as early marker of platelet activation Activated fibrinogen receptor as late marker of platelet activation
Change of in vitro bleeding time using the Platelet Function Analyzer (PFA-100) | At 2 weeks supplementation
  Using collagen-epinephrine coated cartridges Using collagen-adenosine diphosphate coated cartridges
Change of coagulation marker assessed as fibrinogen levels in plasma | At 2 weeks supplementation
  Using semi-automated coagulometer using fibrinogen assay according to Clauss method

SECONDARY OUTCOMES:
Change in light transmission aggregometry of platelet rich plasma induced by collagen and arachidonic acid | At 2 weeks supplementation
  Using a Helena Platelet Aggregation Chromogenic Kinetics System-4 (PACKS-4) light transmission aggregometer
Change in plasma levels of von Willebrand factor (vWF), soluble ICAM (s-ICAM) and soluble P-selectin (sP-selectin) as markers of endothelial activation | At 2 weeks supplementation
  Using enzyme-linked immunoabsorbent assay (ELISA) in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Baukje De Roos, PhD, Principal Investigator — Univeristy of Aberdeen
Locations (1):
- Rowett Institute of Nutrition and Health, Aberdeen, Scotland, United Kingdom

REFERENCES:
- [Background] Benito P, Nelson GJ, Kelley DS, Bartolini G, Schmidt PC, Simon V. The effect of conjugated linoleic acid on platelet function, platelet fatty acid composition, and blood coagulation in humans. Lipids. 2001 Mar;36(3):221-7. doi: 10.1007/s11745-001-0711-y. PMID 11337976
- [Background] Bhattacharya A, Banu J, Rahman M, Causey J, Fernandes G. Biological effects of conjugated linoleic acids in health and disease. J Nutr Biochem. 2006 Dec;17(12):789-810. doi: 10.1016/j.jnutbio.2006.02.009. Epub 2006 May 2. PMID 16650752
- [Background] Malpuech-Brugere C, Verboeket-van de Venne WP, Mensink RP, Arnal MA, Morio B, Brandolini M, Saebo A, Lassel TS, Chardigny JM, Sebedio JL, Beaufrere B. Effects of two conjugated linoleic Acid isomers on body fat mass in overweight humans. Obes Res. 2004 Apr;12(4):591-8. doi: 10.1038/oby.2004.68. PMID 15090626
- [Background] Zhila VV, Shodmonova ZR, Rublevskii VP, Chernenko PS. [High resection of the left testicular vein and ligation of the internal iliac artery using a retroperitoneoscope]. Klin Khir (1962). 1991;(5):49-51. Russian. PMID 1875623
- [Background] Moloney F, Yeow TP, Mullen A, Nolan JJ, Roche HM. Conjugated linoleic acid supplementation, insulin sensitivity, and lipoprotein metabolism in patients with type 2 diabetes mellitus. Am J Clin Nutr. 2004 Oct;80(4):887-95. doi: 10.1093/ajcn/80.4.887. PMID 15447895
- [Background] Brewerton TD, Murphy DL, Lesem MD, Brandt HA, Jimerson DC. Headache responses following m-chlorophenylpiperazine in bulimics and controls. Headache. 1992 May;32(5):217-22. doi: 10.1111/j.1526-4610.1992.hed3205217.x. PMID 1628957
- [Background] Noone EJ, Roche HM, Nugent AP, Gibney MJ. The effect of dietary supplementation using isomeric blends of conjugated linoleic acid on lipid metabolism in healthy human subjects. Br J Nutr. 2002 Sep;88(3):243-51. doi: 10.1079/BJN2002615. PMID 12207834
- [Background] Riserus U, Vessby B, Arnlov J, Basu S. Effects of cis-9,trans-11 conjugated linoleic acid supplementation on insulin sensitivity, lipid peroxidation, and proinflammatory markers in obese men. Am J Clin Nutr. 2004 Aug;80(2):279-83. doi: 10.1093/ajcn/80.2.279. PMID 15277146
- [Background] Riserus U, Vessby B, Arner P, Zethelius B. Supplementation with trans10cis12-conjugated linoleic acid induces hyperproinsulinaemia in obese men: close association with impaired insulin sensitivity. Diabetologia. 2004 Jun;47(6):1016-9. doi: 10.1007/s00125-004-1421-8. Epub 2004 May 28. PMID 15168020
- [Background] Riserus U, Basu S, Jovinge S, Fredrikson GN, Arnlov J, Vessby B. Supplementation with conjugated linoleic acid causes isomer-dependent oxidative stress and elevated C-reactive protein: a potential link to fatty acid-induced insulin resistance. Circulation. 2002 Oct 8;106(15):1925-9. doi: 10.1161/01.cir.0000033589.15413.48. PMID 12370214
- [Background] Riserus U, Arner P, Brismar K, Vessby B. Treatment with dietary trans10cis12 conjugated linoleic acid causes isomer-specific insulin resistance in obese men with the metabolic syndrome. Diabetes Care. 2002 Sep;25(9):1516-21. doi: 10.2337/diacare.25.9.1516. PMID 12196420
- [Background] Tholstrup T, Raff M, Straarup EM, Lund P, Basu S, Bruun JM. An oil mixture with trans-10, cis-12 conjugated linoleic acid increases markers of inflammation and in vivo lipid peroxidation compared with cis-9, trans-11 conjugated linoleic acid in postmenopausal women. J Nutr. 2008 Aug;138(8):1445-51. doi: 10.1093/jn/138.8.1445. PMID 18641189
- [Background] Tricon S, Burdge GC, Kew S, Banerjee T, Russell JJ, Jones EL, Grimble RF, Williams CM, Yaqoob P, Calder PC. Opposing effects of cis-9,trans-11 and trans-10,cis-12 conjugated linoleic acid on blood lipids in healthy humans. Am J Clin Nutr. 2004 Sep;80(3):614-20. doi: 10.1093/ajcn/80.3.614. PMID 15321800
- [Background] Truitt A, McNeill G, Vanderhoek JY. Antiplatelet effects of conjugated linoleic acid isomers. Biochim Biophys Acta. 1999 May 18;1438(2):239-46. doi: 10.1016/s1388-1981(99)00055-4. PMID 10320806
- [Derived] Bachmair EM, Wood SG, Keizer HG, Horgan GW, Ford I, de Roos B. Supplementation with a 9c,11t-rich conjugated linoleic acid blend shows no clear inhibitory effects on platelet function in healthy subjects at low and moderate cardiovascular risk: a randomized controlled trial. Mol Nutr Food Res. 2015 Apr;59(4):741-50. doi: 10.1002/mnfr.201400495. Epub 2015 Feb 23. PMID 25641922